CLINICAL TRIAL: NCT04998526
Title: The Effect of Local Cold Application on Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Collaborators: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, YAVUZ ÜREN, PhD Student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yavuztez
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
Keywords: Cold application; Headache; Heart rate; Nursing
MeSH Terms: conditions — Hypertension; Headache

STUDY DESIGN:
Intervention Model Description: This study, which is planned as a randomized controlled and experimental study, will be conducted with type 2 (systolic blood pressure between 160 and 179 mmHg, diastolic blood pressure between 100 and 109 mmHg) essential hypertension patients who refer to Van Yüzüncü Yıl University Dursun Odabaş Medical Centre Emergency Service. The patients will be distributed as 24 in experimental group, 24 in placebo group and 24 in control group based on block randomization (gender and age) method and a total of 72 patients will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): After routine drug treatment is given to hypertension patients, the cold gel pack will be applied to the nape for 3 minutes.
  Interventions: Other: Experimental group
- Placebo group (Placebo Comparator): After routine drug therapy is given to hypertension patients, the gel pack kept at room temperature will be applied to the nape for 3 minutes.
  Interventions: Other: Placebo group
- Control group (No Intervention): Routine drug treatment will be given to hypertension patients and no application will be made.

INTERVENTIONS:
Other: Experimental group — The cold gel pack will be applied to the nape.
  Other Names: Cold application
  Arms: Experimental group
Other: Placebo group — The gel pack kept at room temperature will be applied to the nape.
  Arms: Placebo group

SUMMARY:
This study will be conducted to evaluate the effect of local cold application to the nape of the neck on systolic blood pressure, diastolic blood pressure, heart rate, heart rate pressure and headache.

DETAILED DESCRIPTION:
Aim: This study will be conducted to evaluate the effect of local cold application to the nape of the neck on systolic blood pressure, diastolic blood pressure, heart rate, heart rate pressure and headache.

Material and method: This study, which is planned as a randomized controlled and experimental study, will be conducted with type 2 (systolic blood pressure between 160 and 179 mmHg, diastolic blood pressure between 100 and 109 mmHg) essential hypertension patients who refer to Van Yüzüncü Yıl University Dursun Odabaş Medical Centre Emergency Service. The patients will be distributed as 24 in experimental group, 24 in placebo group and 24 in control group based on block randomization (gender and age) method and a total of 72 patients will be included. Patient information form, blood pressure and heart rate monitoring form and VAS pain scale will be used to collect study data. Patients in all groups will be measured in 90 minutes for a total of 8 times, as pre-test (pre-application) and post-test (minutes 3, 10, 15, 20, 30, 60 and 90). After routine medication therapy is given to all three groups, the cold gel pack which has been kept at least for four hours in the freezer will be applied to the nape of the patients in the experimental group, while gel pack at room temperature will be applied to the placebo group and no application will be made to the control group. Variance analysis, Friedman analysis, t test, Wilcoxon test and Kruskal Wallis analysis will be used in data assessment.

ELIGIBILITY:
Inclusion Criteria:

* 25 mg sublingual ACE inhibitor given as a treatment protocol,
* No wound on the nape,
* Does not develop cold intolerance,
* Not taking any hypertension medication and pain medication in the last 6 hours,
* Without heart diseases, peripheral arterial circulation disorders, sensory disorders and edema,
* Not pregnant,
* Agreeing to participate in the study,
* Essential hypertension patients with systolic blood pressure 160 - 179 mmHg, diastolic blood pressure 100 - 109 mmHg.

Exclusion Criteria:

* Developing cold intolerance,
* Changes in the treatment regimen,
* Panic attack, allergic reaction and any similar situation develops,
* Those who want to withdraw from the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 90 minute
  Lowering blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: YAVUZ ÜREN, PhD Student, Principal Investigator — Ataturk University; EMİNE KIYAK, Prof.Dr., Study Chair — Ataturk University; SEVDEGÜL BİLVANİSİ, Prof.Dr., Study Chair — Yuzuncu Yil University
Locations (1):
- Van Yüzüncü Yıl University Dursun Odabaş Medical Centre Emergency Service, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No